CLINICAL TRIAL: NCT03541707
Title: Evaluation of the H1-Coil TMS- Double Blind Placebo Controlled Study in Adolescent Patients Suffering From Major Depression.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Yuval Bloch, Head of Child and Adolescent Outpatient clinic and Research Unit, Shalvata Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0020-17 SHA
Record Dates: First submitted 2018-04-16; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Depression
Keywords: TMS; EEG; Depression; adolescents
MeSH Terms: conditions — Depression | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: Fifty-two adolescent patients suffering from major depression that are still severely ill after at least one psychological treatment and at least 2 adequate treatments knowledge of patient or doctor who receives the active therapy. Patients will be evaluated for efficacy, side effects, and cognitive performance. Brain waves (using EEG) will be monitored to see if they can predict who will respond to deep TMS.with medications, will be recruited. After the informed consent of guardians and patients, a systematic clinical evaluation with the aid of appropriate questionnaires will be performed. Patients will be allocated in a randomized double blind placebo controlled manner to dTMS or Sham treatments for about half an hour per day over 20 consecutive working days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be allocated, based on chance, to receive active therapy or a "as if" stimulation, with no knowledge of patient or therapist who receives the active therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Therapy (Active Comparator)
  Interventions: Device: Deep TMS Brainsway's H coil
- "As if" Stimulation (Sham Comparator)
  Interventions: Device: Deep TMS Brainsway's H coil

INTERVENTIONS:
Device: Deep TMS Brainsway's H coil — During the treatment trial period all subjects will receive the following dose of TMS: 18 Hz, at 100% RMT, 2 sec pulse train, 20 second inter-train interval, 80 trains, for a total of 57,600 pulses over the complete treatment course. In the placebo group a state of the art sham procedure will be used- the coil is programed to produce the noise and local sensation but with no activation.
  EEG Recording is done with and without an acoustic oddball trigger, in order to have both resting state and event related recordings. The evaluation takes approximately 5 minutes.
  Other Names: EEG (MindWave of NeuroSky LTD)

SUMMARY:
This study is a randomized double blind placebo controlled EEG monitored study of deep rTMS treatment to treat adolescent depression.

The present study is the first well controlled study to examine the possible clinical utility of deep TMS to treat a severe and life threatening disorder- depression, among adolescents.

Patients will be allocated, based on chance, to receive active therapy or a "as if" stimulation, with no knowledge of patient or therapist who receives the active therapy. In addition, a simple and feasible monitoring of brain waves (EEG) will be conducted. This addition will enable us to evaluate the possibility to use biological markers to predict the course of therapy.

Our hypothesis is that 1. patients receiving the active therapy will improve significantly more than those who received the "as if" treatment. 2. There will be no significant side effects. 3. The brain waves (as measured by the EEG) will predict treatment response.

DETAILED DESCRIPTION:
Adolescent depression is a severe disorder affecting 5-8% of adolescents. It is a major risk factor for adolescent suicide-one of the 3 most common reasons for death in this age group. It carries with it a heavy burden of harsh comorbidities such as substance abuse, and behavioral problems[1, 2].

The first line treatment of moderate or severe illness includes pharmacotherapy with serotonin reuptake inhibitors (SSRIs) such as fluoxetine, in combination with psychotherapy. However, more than 30% of the patients do not achieve remission (defined as minimal or no symptoms) despite treatment with a combined intervention [3]. In adolescents there is some evidence that as a second line, switching to another SSRI combined with cognitive behavioral therapy (CBT) can be useful [4]. There is no evidence to what should be the third line in therapy. Early intervention in the course of a disease is expected to protect from the grave long term sequelae[9], but in treating adolescent depression our therapeutic tools are extremely limited[10].

There is a necessity to advance our evidence based interventions to treat treatments resistant adolescent depression.

Hypoactivity in the left dorsolateral prefrontal cortex (DLPC) is a key finding in brain imaging of depression[11]. Repetitive transcranial magnetic stimulation (rTMS) is a therapeutic procedure in which a magnetic coil that generates recurrent pulsatile magnetic fields from a rapidly oscillating electrical current is placed on the scalp, to induce recurrent electrical currents in the brain. High frequency rTMS causes activation of the affected brain regions and networks. This is the suggested mechanism of the antidepressant effect of high frequency rTMS to the left DLPC in depression[12]. Recent advances in custom coil technology led to the development of H coils that support stimulation of deeper, limbic structures[13]. Due to the accumulating knowledge on safety and efficacy in adult depression both the custom rTMS and the "deep" H coil TMS are approved (FDA and Israeli ministry of health), for clinical (not just research) use [12, 14-16]. In a large multicenter study of the H1 coil to treat adult depression there were minimal side effects and a large effect size of 0.78 was reported, strengthening the promise of this mode of therapy [5].

The field of brain stimulation and specifically TMS is based on the concept of neuroplasticity, the ability of repeated stimulations to cause a longer lasting neuronal change. In this respect the adolescent developing brain is a period of opportunity for such changes[17, 18] To date, there are no randomized placebo controlled studies on rTMS to treat adolescents suffering from depression, although reports support the safety of rTMS in treating adolescents. Recently, there was a report of a self-limited convulsion in an adolescent treated with deep rTMS at 120% motor threshold-strengthening the necessity for well-structured studies in the field[23].

Studying biomarkers holds the promise for translating neuroscientific understandings to the clinical practice of adolescent depression[24]. In order to be useful a biomarker has to be discriminative (between responder vs non responder for example), to reflect a pathophysiological process, but last and not least it is important that it will be accessible for use[25, 26]. This explains the evolving interest in using electroencephalography (EEG) findings to study depression and monitor the course of therapy[27, 28]. Imaging and electrophysiological studies support the importance of the interplay between the attentional and default networks as a marker of the disease course[29, 30]. In a recent study our group cooperated in a study of a new simple EEG technique, that by using repeated simple attentional EEG measures was able to predict treatment response in a heterogeneous group of adult depressed patients[31]. These safe and simple markers were never studied in adolescent depression.

The present research is a randomized double blind placebo controlled EEG monitored study of deep rTMS treatment to treat adolescent depression.

Research goals and expected significance:

1. To study the efficacy and safety of deep rTMS to treat treatments resistant adolescent depression. As there are no well controlled studies of rTMS to treat adolescent depression, the possibility to evaluate a new therapeutic tool for this severe, life threatening disease has immense clinical value. Since this technique is based on evolving neuroscientific understandings, it holds promise for advancing our understanding of adolescent depression.
2. To evaluate a potential pragmatic EEG measure to predict and monitor therapeutic outcome. Since the effect of deep rTMS on the developing brain of the depressed adolescent has a potential for both therapy and side effects, early prediction of the effect is crucial. The potential of having biomarkers to complement clinical and subjective evaluations is of paramount importance for personalizing, objectively monitoring therapy to treat adolescent depression.

Methods:

Subjects: Fifty-two adolescents (age: 14-18y) suffering from treatment resistant depression will be recruited from "Shalvata mental health center" in patient ward, and outpatient facilities. Sample size calculation was based on the effect size of 0.78 found in the adult depression study[5]. The Shalvata Mental Health Center serves a large catchment area, and the investigators are experienced in recruiting depressed adolescent patients to rTMS studies [20, 21, 33]. Participation will be based on the following criteria:

Devices:

Deep TMS Brainsway's H coil, and deep TMS are registered in Israel for clinical use to treat depression in adults. Our center has gained years of experience in studies with this system[5, 16, 32, 37]. Deep TMS treatments will be carried out by a technician (trained and approved by the manufacturer) that will remain in the treatment room during the entire procedure. In addition, a physician will be available on-call within the hospital grounds.

At the beginning of the trial individual motor threshold (MT) will be measured by placing the assigned coil above the hand area of the motor cortex. Patients will receive stimulations over the prefrontal cortex, 6 cms anterior to the 'hot spot' for stimulation of the abductor policies brevis in the hand area. Each deep TMS treatment will be conducted as follows: Before starting each treatment, patients will be instructed to insert earplugs to lessen any possible adverse effect on hearing. Twice a week, the MT will be measured by delivering single stimulations to the motor cortex. The MT is measured by gradually increasing the intensity. This is done by using the single pulse mode and applying one pulse every 5 secs, i.e. 0.2 Hertz. The electrical activity in abductor pollicis brevis is then recorded using surface electrodes. Threshold is defined as the lowest intensity of stimulation able to produce motor evoked potentials of at least 50µV in 5 of 10 trials. After defining the motor threshold, the same intensity will be used in following treatments until the next threshold examination. The coil will be positioned 6 cm anterior to the hot spot (according to clinical judgment of the physician in charge, The reference point could move 5 anterior to the hot spot) and an dTMS session will be performed at 100% of the motor threshold, for safety the investigatores lowered the 120% threshold used with adult depressed subjects.

During the treatment trial period all subjects will receive the following dose of TMS: 18 Hz, at 100% RMT, 2 sec pulse train, 20 second inter-train interval, 80 trains, for a total of 57,600 pulses over the complete treatment course. In the placebo group a state of the art sham procedure will be used- the coil is programed to produce the noise and local sensation but with no activation[38].

MindWave of NeuroSky LTD This is an simple and approved EEG system, that enables us to produce off line with the technology of Brain marc a valuable marker related to attention[39]. The recording will be performed by a trained technician and carries no danger and minimal inconvenience. Recording is done with and without an acoustic oddball trigger, in order to have both resting state and event related recordings. The evaluation takes approximately 5 minutes. The data are transported as anonymous signals to a secured cloud. Our group has had fruitful experience with working with this system with depressed patients[31].

Cognitive assessment:

Computerized Neuropsychological Battery (Penn CNP) In studying innovative treatments for adolescent depression cognitive and affective assessments are extremely important. Depression has state and trait effects on cognitive abilities including attention and working memory[40, 41]. Since possible effect on memory is a central concern with the use of electroconvulsive therapy considered by some the prototype of brain stimulation techniques monitoring cognitive functions especially in an adolescent brain stimulation (TMS) study is crucial[42, 43]. The web-based Computerized Neuropsychological Battery (Penn CNP) of the Brain Behavior Laboratory at the University of Pennsylvania offers a range of probes of human neuropsychological functioning (www. penncnp.med.upenn.edu). It was designed for neuropsychological measurement of major cognitive domains. PennCNP has granted us permission to use the WenCNP battery after assurance that our study is held in research institutions with IRB support, under the direction of accredited research faculty members or students. The WebCNP is administered using clickable icons on desktop or laptop computers, in a fixed order. An Applescript® routine is used to collect participant IDs and basic demographic information and to present the tests in a prescribed order. The test administrator reads instructions for each test and observes as the participant performs the tests. Administrating the tests in a standard fashion fostering optimal performance without aiding the participant is required. The test administrator provides a status code and comments regarding the validity of collected data. The results are uploaded to a data repository using an automated script, and scored using a program written in the Python programming language. For each domain, accuracy (number of correct responses) and speed (response time for correct answers) are computed. Full battery completion takes approximately 1 hour. Each test begins with a practice module, to assure understanding of the instructions. The tasks in the battery include the following: Motor Praxis Test, The Penn Face Memory Test, Short Visual Object Learning Test, Short Penn continuous performance task (CPT), Short Letter N-Back Task, Penn Facial Memory Test- Delayed, Memory Short Visual Object Learning Test - Delay, Penn Emotion Recognition Faces 40, The Penn Conditional Exclusion Test, The Penn Word Memory Test, Penn Emotion Discrimination Task, Short Penn Computerized Tapping Task, Penn Matrix Analysis Test, Penn Facial Age discrimination, Variable Short Penn Line Orientation Test (34).

Clinical Questionnaires:

The development and well-being assessment (DAWBA). Is a commonly used structured interview intended to improve diagnostic reliability [34].

CGI - Clinical Global Impression: CGI is a commonly used tool for assessing the severity of the patient's depression. It uses 7 levels, ranging from normal to severely ill[36]. It is important to note that this is a course but extremely relevant measure used in some of the most influential studies on treating adolescent depression[3].

Child depression rating scale (CDRS) Is a well validated structured assessment of adolescent depression, using questions relevant to this age group[35].

Quick Inventory of Depressive Symptomatology (QIDS-SR). This is self-report commonly used in studying and monitoring depression in different age groups[44].

Suicidal ideation questionnaire (SIQ). This evaluation tool has shown reliability and validity in assessing and monitoring the severity of suicidal ideation[45].

The screen for child anxiety and related emotional disorders (SCARED). This is a brief and well established questionnaire that helps evaluate anxiety, highly relevant measure in depressed adolescents[46].

Experimental design:

After a brief presentation and screen eligible patients and their guardians will be invited to complete the informed consent process.

Visit 1-pretreatment evaluation:

Will include a physical and psychiatric evaluation completed with the DAWBA[34] interview, the CDRS[35] to evaluate depression severity, the suicidal ideation questionnaire (SIQ)[45] and the CGI[36]. Patients will complete a demographic questionnaire, QIDS [44], the screen for child anxiety and related emotional disorders SCARED[46]. In addition patients will go through a cognitive evaluation using the Penn Web-Based Computerized Neurocognitive Battery (WebCNP)[47]. On this visit the first EEG evaluation will be performed[31].

After the pretreatment visit patients will be blindly randomized to active or sham procedure.

Visit 2-21 On visit 2 treatment threshold will be determined. For the next 4 weeks patients will have a daily treatment (sham or active) session on each working day (5 days a week). Before and after each treatment patients will be asked about their general condition, mood, suicidal thoughts and side effects from the treatment. Before each therapy day an EEG monitoring will be performed.

On visits 2, 7, 12, 17 and 21 (the first visit of every week, and the last session), patients will complete the clinical evaluation using the questionnaires detailed in the screen, and repeat the EEG assessment after therapy.

Follow up visits, visits 22-24:

After a week (visit 22), a month (visit 23) and two months (visit 24) patients will repeat the more detailed evaluation as on the weekly visits. On visit 22 the cognitive evaluation done in the screen will be repeated.

Study Duration The anticipated enrollment rate is 2-3 per month. Therefore, approximately 20 months will be required to enroll 52 subjects. The protocol duration for each subject is 4 weeks, followed by 8 weeks for the 2 follow-up visits; therefore the total study duration including data processing is expected to be approximately 24 months. After an ethical consultation it has been decided that patients who were in the sham group, at the end of the blinding will be able to receive active therapy.

Monitoring of Subjects and Criteria for Withdrawal During the entire study, the subjects will be under the direct monitoring of the principal investigator. Any adverse effect or subjective disturbance will be immediately recorded and responded to. If subjects are not cooperative, they may be withdrawn by the investigators. Subjects or parents wishing to withdraw at any time would be able to do so without prejudice. Subjects whose condition is deteriorating as expressed by a 15% rise or more in the clinical questionnaires during the study period with no known emotional trigger (such as a family or romantic crisis) will discontinue therapy.

Subject that completed 16 treatments or more, within 6 weeks, will be considered as a subject who completed the study trail.

ELIGIBILITY:
Inclusion Criteria:

* Age: 14-18 years.
* Diagnosed as suffering from major depression by two senior child and adolescent psychiatrist according to DSM 5 criteria, and validated with the development and well-being assessment (DAWBA) interview[34].
* Severe depression as assessed by the child depression rating scale (CDRS)[35] of 40 or more, and the clinical global impression scale (CGI)[36] of 4 or more.
* They have had at least 2 antidepressant drug trials of at least 5 weeks (or 3 drug trials if trials were discontinued earlier due to intolerance), beyond psychotherapy.
* They scored negative on all TMS safety questionnaire.
* There was no change in pharmacotherapy in the past 3 weeks.
* Both patients and guardians have given an informed consent.
* Patients are under continued clinical monitoring.

Exclusion Criteria:

* Patients suffering from schizophrenia.
* Present or history of any general medical or neurological significant disorder including: epilepsies, hypertension, head injuries or neurosurgery, migraine, and hearing loss.
* Substance abuse in the past 2 weeks.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
For efficacy, improvement in the CGI is the primary outcome measure. | 24 months
  Efficacy will be examined by the improvement in Clinical global Impression(CGI).
For safety, severe side effects are the primary outcome measure. | 24 months
  Safety will be examined by Incidence of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
cognitive changes in response to the treatment | 24 months
  As measured by cognitive evaluation using the Penn Web-Based Computerized Neurocognitive Battery (WebCNP)

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata Mental health Center, Hod HaSharon, Israel

IPD SHARING:
Plan to Share IPD: Undecided